CLINICAL TRIAL: NCT00687713
Title: Phase 2, Double-Blind, Placebo-Controlled Trial of Bupropion for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDS Bupropion Meth 0001
Record Dates: First submitted 2008-05-29; First posted 2008-06-02 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Active Comparator): Subjects will receive bupropion 150 mg tablet for 3 days then twice daily, for 12 weeks until dose taper during the last 3 days of week 12 at 150 mg per day.
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Subjects will receive a matched bupropion placebo 150 mg tablet for 3 days then twice daily, for 12 weeks until dose taper during the last 3 days of week 12 at 150 mg per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion — 150mg for the first 3 days of dosing. Increased to 150 mg b.i.d until taper.
  Arms: Bupropion
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is to assess the efficacy of bupropion in reducing methamphetamine use in subjects with methamphetamine dependence who report using methamphetamine 29 or less days during the 30 days prior to the start of signing consent.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy of bupropion in reducing methamphetamine use in subjects with methamphetamine dependence who report using methamphetamine 29 or less days during the 30 days prior to signing consent. Secondary objectives included but were not limited to: assessing the success or failure to achieve abstinence (confirmed by at least two methamphetaminenegative urines and no methamphetamine-positive urines) each week during the last two weeks (Weeks 11 and 12) for subjects using methamphetamine 18 or less days during the 30 days prior to signing consent, assessing the safety of bupropion in this study population, assessing other measures of efficacy of bupropion in reducing methamphetamine use or craving, and other psychological assessments of methamphetamine dependence.

It is hypothesized that bupropion, compared to placebo, would be associated with an increase in the proportion of subjects who achieved abstinence (confirmed by at least two methamphetamine-negative urines and no methamphetaminepositive urines) each week during the last two weeks (Weeks 11 and 12) for non-daily users.

ELIGIBILITY:
Inclusion Criteria:

* Must have a DSM-IV diagnosis of methamphetamine dependence as determined by MINI
* Must have at least 1 amphetamine or methamphetamine positive urine specimen after the start of screening and before randomization or provide information to verify recent use if a positive urine sample can't be obtained
* Must report using methamphetamine for 29 days or less during the 30 day period prior signing consent using the timeline follow-back method
* Must be willing and able to comply with study procedures
* Must be able to verbalize and understand consent forms and provide written informed consent
* Must be seeking treatment for methamphetamine dependence

Exclusion Criteria:

* Please contact study site for more information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jurij Mojsiak, Study Chair — National Institute on Drug Abuse (NIDA)
Locations (12):
- United States (12):
  - UCLA Integrated Substance Abuse Program, Los Angeles, California
  - South Bay Treatment Center, San Diego, California
  - Addiction and Pharmacology Research Laboratory, San Francisco, California
  - Friends Research Institute, Torrance, California
  - Matrix Institute, Woodland Hills, California
  - Pacific Addiction Research Center - U of Hawaii, Honolulu, Hawaii
  - Iowa Luther Hospital, Des Moines, Iowa
  - U of Kansas Medical Center, Kansas City, Missouri
  - New York University, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science At San Antonio, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson AL, Li SH, Markova D, Holmes TH, Chiang N, Kahn R, Campbell J, Dickerson DL, Galloway GP, Haning W, Roache JD, Stock C, Elkashef AM. Bupropion for the treatment of methamphetamine dependence in non-daily users: a randomized, double-blind, placebo-controlled trial. Drug Alcohol Depend. 2015 May 1;150:170-4. doi: 10.1016/j.drugalcdep.2015.01.036. Epub 2015 Feb 7. PMID 25818061

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion: Subjects received bupropion 150 mg tablet for 3 days then twice daily, for 12 weeks until dose taper during the last 3 days of week 12 at 150 mg per day.
  Bupropion: 150mg for the first 3 days of dosing. Increased to 150 mg b.i.d until taper.
- Placebo: Subjects received a matched bupropion placebo 150 mg tablet for 3 days then twice daily, for 12 weeks until dose taper during the last 3 days of week 12 at 150 mg per day.
  Placebo: Placebo
Period: Overall Study
Arm/Group | Bupropion | Placebo
Started | 100 | 104
Completed | 68 | 64
Not Completed | 32 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion | Placebo | Total
Number analyzed (Participants) | 100 | 104 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 104 | 204
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 63 | 69 | 132
Region of Enrollment [Number; unit: participants]
  United States | 100 | 105 | 205

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Showing Abstinence
Description: The primary efficacy outcome measure was a measurement of treatment success or failure, where a subject who successfully achieved two weeks of abstinence during the last two weeks of investigational product dosing (Weeks 11 and 12) was scored as a success.
Time Frame: Weeks 11 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 100 | 104
Participants | 14 | 20

2. Secondary Outcome: Treatment Success Among Subjects With 18 or Less Days of Methamphetamine Use
Description: The study population for this outcome measure is defined as those participants with methamphetamine dependence who report using methamphetamine 18 or less days during the 30 days prior to signing consent.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bupropion | Placebo
Number analyzed (Participants) | 100 | 104
Participants | 65 | 76

ADVERSE EVENTS:
Arm/Group | Bupropion | Placebo
Serious Adverse Events (participants affected / at risk) | 1/100 | 3/104
Other Adverse Events (participants affected / at risk) | 83/100 | 93/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion (N=100) | Placebo (N=104)
Gastric bypass (Gastrointestinal disorders) | 1 | 3 — Subject underwent elective gastric bypass surgery without complication. Was hospitalized and discharged 3 days later. Severity was moderate. Event was unexpected and definitely not related to study drug. She is recovered and continued in the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion (N=100) | Placebo (N=104)
Nausea (Gastrointestinal disorders) | 9 (14) | 23 (27)
Headache (Nervous system disorders) | 37 (68) | 43 (88)
Nasopharyngitis (Infections and infestations) | 4 (5) | 12 (12)
Back Pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No